CLINICAL TRIAL: NCT05048680
Title: Effect of Hypoxic Conditioning on Cerebrovascular Health in the Elderly
Acronym: HYPOXAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 38RC20.460
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Hypoxia; Cerebral Hypoxia; Brain Diseases; Exercise; Aging; Cognitive Decline; Healthy Aging
MeSH Terms: conditions — Hypoxia; Hypoxia, Brain; Brain Diseases; Motor Activity; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind (participant and research team) study in relation to the gas being delivered (normoxic or hypoxic mixture) during intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hypoxia - Rest (Experimental): Sessions of intermittent hypoxia at rest; 3 sessions/week; 8 weeks. To be compared with the placebo (normoxia) group at rest.
  Interventions: Procedure: Hypoxia and/or Exercise
- Normoxia - Rest (Placebo Comparator): Sessions of normoxia at rest; 3 sessions/week; 8 weeks.
  Interventions: Procedure: Hypoxia and/or Exercise
- Hypoxia - Exercise (Experimental): Sessions of exercise training under hypoxia; 3 sessions/week; 8 weeks. To be compared with the placebo (exercise under normoxia) group.
  Interventions: Procedure: Hypoxia and/or Exercise
- Normoxia - Exercise (Active Comparator): Sessions of exercise training under hypoxia; 3 sessions/week; 8 weeks.
  Interventions: Procedure: Hypoxia and/or Exercise

INTERVENTIONS:
Procedure: Hypoxia and/or Exercise — Hypoxia at rest versus normoxia at rest; Hypoxia during exercise versus Normoxia during exercise.

SUMMARY:
In line with the ever-growing aging of Western populations, the development of preventive strategies to slow down the effects of aging on cardiovascular health represents a major challenge in order to preserve functional capacities and a sufficient quality of life in the elderly. The alteration of vascular function (at the cerebral and systemic level) with aging is an important feature in the clinical picture including a decrease in physical and cognitive capacities. Although physical activity is recognized as an essential means of combating the effects of aging, optimizing its effects by defining the most effective strategies of practice remains a key objective. Offering alternative interventions to exercise training is also necessary for people who are unwilling or unable to engage in a physical activity program. In this context, hypoxic conditioning, alone or in conjunction with rehabilitative exercise training, is a new therapeutic modality with strong preclinical validity, in particular from a cardiovascular standpoint, and used in other pathologies to improve cardiovascular function and exercise performance and quality of life. Our aim is, therefore, to investigate the effect of hypoxic conditioning (alone or in conjunction with exercise training) on cerebrovascular health in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 80 years of age;
* Being physically inactive (less than 150 min/week of moderate to intense physical activity);
* No chronic cardiovascular, respiratory, metabolic or neuromuscular disease counterindicating an exercise training or hypoxic conditioning program;
* Health coverage;
* Being able to provide written fully informed consent.

Exclusion Criteria:

* Body-mass index >30 kg/m2;
* Smoking (> cigarettes/day);
* Alcohol use (> 10g/day);
* Mental disorder or history of mental disorder;
* Beta-blockade treatment;
* Inability or refusal to provide informed consent;
* No health coverage
* People exceeding the annual ceiling of allowances received as a result of their participation in other clinical trials;
* People deprived of freedom by judicial or administrative decision;
* People subject to legal protection, who cannot be included in clinical trials.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Middle cerebral artery flow velocity | Before intervention; right after intervention; 2 months after intervention
  Changes in middle cerebral artery flow velocity in response to hypercapnia (5% CO2)

SECONDARY OUTCOMES:
Peak oxygen uptake | Before intervention; right after intervention; 2 months after intervention
  Peak oxygen uptake during a cardiopulmonary exercise test
Flow-mediated dilation | Before intervention; right after intervention; 2 months after intervention
  Flow-mediated dilation in response to ischemia-reperfusion of the brachial artery
Blood pressure | Before intervention; right after intervention; 2 months after intervention
  24h (systolic, diastolic and mean) blood pressure assessment
Sleep | Before intervention; right after intervention; 2 months after intervention
  Sleep features assessed by polygraphy
Cognitive function | Before intervention; right after intervention; 2 months after intervention
  Cognitive function assessed by the Montreal Cognitive Assessment questionnaire
Health-related quality of life | Before intervention; right after intervention; 2 months after intervention
  Health-related quality of life assessed by the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Doutreleau, MD, PhD, Principal Investigator — CHU Grenoble Alpes, Grenoble Alpes University
Locations (1):
- CHU Grenoble Alpes, La Tronche, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No
No plan at this point in time.